CLINICAL TRIAL: NCT01583361
Title: Phase III, Randomized, Multicenter, Controlled Evaluation of S-1 and Oxaliplatin as Neoadjuvant Chemotherapy for Advanced Gastric Cancer Patients
Brief Title: SOX Regimen as Neoadjuvant Chemotherapy for AJCC Stage II-III Gastric Cancer
Acronym: RESONANCE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lin Chen (Other)
Responsible Party: Sponsor-Investigator, Lin Chen, Chief of GI Surgeon, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCHEN-PLAGH
Record Dates: First submitted 2012-04-04; First posted 2012-04-24 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Gastric Adenocarcinoma
Keywords: two arms; D2 lymphadenectomy; chemotherapy before and after surgery; disease free survival

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A:Neoadjuvant sox (Experimental): Patients in arm a will receive (N=2-4) cycles of neoadjuvant SOX first, and then standard gastrectomy with D2 lymphadenectomy, and (8-N) cycles of adjuvant SOX adjuvant chemotherapy.
  Interventions: Drug: Oxaliplatin+S-1
- Arm B:Adjuvant SOX (Active Comparator): Patients in arm B will receive standard gastrectomy with D2 Lymphadenectomy first, and 8 cycles of adjuvant SOX later.
  Interventions: Drug: Adjuvant Oxaliplatin/S-1（SOX）

INTERVENTIONS:
Drug: Oxaliplatin+S-1 — S-1: 40~60mg bid，po, d1~14 （S-1：BSA <1.25m2, 40mg bid, 1.25m2≤BSA≤1.5m2,50mg bid, BSA>1.5m2, 60mg bid） oxaliplatin：130mg/m2，iv drip for 2h，d1
  Other Names: Oxaliplatin(Sanofi-aventis); S-1(Taiho)
  Arms: Arm A:Neoadjuvant sox
Drug: Adjuvant Oxaliplatin/S-1（SOX） — S-1：40~60mg bid，d1~14 q3W oxaliplatin：130mg/m2，iv drip for 2h，d1,q3W 8 cycles (6 months)
  Other Names: Oxaliplatin(Sanofi-aventis); S-1(Taiho)
  Arms: Arm B:Adjuvant SOX

SUMMARY:
This is a randomized, multicenter, controlled trial to prove efficacy of S-1 and Oxaliplatin as Neoadjuvant Chemotherapy for Advanced Gastric Cancer Patients who undergo D2 gastrectomy.

The primary endpoint is three-year free disease and the second primary includes five-year overall survival, safety and R0 resection rate.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed gastric adenocarcinoma
2. Gastroesophageal junction tumour type II or III(NCCN 2009) can be enrolled
3. All patients must undergo EUS,CT(or PET-CT) and laparoscopy to evaluate tumor stage classification (TNM), and only stage II or III (AJCC 7th) gastric cancer patients can be enrolled
4. planning to undergo gastric cancer D2 surgery after neoadjuvant chemotherapy
5. KPS > 60; ECOG performance status 0-2
6. Life expectancy > 6 months
7. Age: 20 to 75 years
8. No other severe disease and life expectancy less than five years
9. 7 days before enrolled, baseline data should be finished including:

   * Granulocyte count ≥ 1.5×109/L;
   * platelet count ≥ 100×109/L;
   * Hemoglobin ≥ 90g/L;
   * hepatic < 1.5×ULN;
   * total bilirubin ≤ 1.0×ULN;
   * creatinine < 1.5×ULN;
   * PT-INR/PTT < 1.7× ULN
10. Disease had to be measurable by the Response Evaluation Criteria in Solid Tumors (RECIST1.1) criteria
11. Written informed consent and able to comply with the protocol

Exclusion Criteria:

1. Patient cannot undergo surgery or chemotherapy because of other severe disease
2. Be allergic to chemotherapy drugs
3. Patients receiving any chemotherapy or drugs involved in this trial in four weeks before enrolled
4. Patients received cytotoxic chemotherapy, targeted therapy, immunotherapy or radiotherapy for gastric cancer
5. Within the last 5 years in patients with a history of other malignant diseases
6. Pregnant or breast-feeding women
7. Severe heart disease like symptoms of coronary heart disease, New York Heart Association (NYHA) grade II or worse congestive heart failure or cardiac arrhythmia having medications or myocardial infarction within the last 12 months
8. Patients with upper gastrointestinal obstruction or absorption anomaly; patient in obstruction of the Helicobacter pylori failure like effect S-1 to take and absorb
9. Patients with a history of peripheral nerve disease
10. Patients who get organ transplant
11. lack of dihydropyrimidine dehydrogenase (DPD)
12. Infection or other disease failure to control

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 772 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-09 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
disease free survival | three years
  SOX regimen as Neoadjuvant chemotherapy for AJCC II-III gastric cancer patients is superior than postoperative SOX after D2 surgery.Disease free survival is defined as time of surgery to recurrence or death.

SECONDARY OUTCOMES:
response rate | 3 months
  For neoadjuvant chemotherapy patients,response rate will be evaluated according to RECIST 1.1 criteria after at least 2 cycles of SOX chemotherapy.CT scan is required to every patient.
overall survival | five years
  Neoadjuvant chemotherapy of SOX is superior than postoperative SOX after D2 dissection in AJCC II-III gastric cancer patients.Overall survival is defined as the time of randomization to death.
safety | six months
  Number of participants with adverse events related to SOX chemotherapy.All adverse events are from CTCAE 4.0 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang X, Lu C, Wei B, Li S, Li Z, Xue Y, Ye Y, Zhang Z, Sun Y, Liang H, Li K, Zhu L, Zheng Z, Zhou Y, He Y, Li F, Wang X, Liang P, Huang H, Li G, Shen X, Ji J, Tang Y, Xu Z, Chen L; RESONANCE study group. Perioperative versus adjuvant S-1 plus oxaliplatin chemotherapy for stage II/III resectable gastric cancer (RESONANCE): a randomized, open-label, phase 3 trial. J Hematol Oncol. 2024 Apr 8;17(1):17. doi: 10.1186/s13045-024-01536-7. PMID 38589926